CLINICAL TRIAL: NCT03673449
Title: A Pilot Study to Evaluate the Reconstruction of Digital Nerve Defects in Humans Using an Implanted Silk Nerve Guide
Brief Title: Evaluate the Reconstruction of Digital Nerve Defects in Humans Using an Implanted Silk Nerve Guide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Silk Biomaterials srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB_DND-01/2018
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Peripheral Nerve Injury Digital Nerve Hand
Keywords: peripheral nerve injury; nerve guide; silk fibroin; silk; nerve regeneration
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Intervention Model Description: Open Label Monocentre Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SilkBridge treatment (Experimental): Surgery for digital nerve reconstruction with SilkBridge
  Interventions: Device: SilkBridge

INTERVENTIONS:
Device: SilkBridge — SilkBridge is a biocompatible silk fibroin-based scaffold, which recruits the patients' own cells to remodel or regenerate the nerve, without pre-seeding of the scaffold nor biological/chemical treatments.

SUMMARY:
The goal of this study is to ascertain the feasibility and safety of the procedure using SilkBridge - a biocompatible silk fibroin-based scaffold - for the regeneration of sensory nerve fibres and follow it up together with the reinnervation of the target organs (sensory receptors in the skin).

DETAILED DESCRIPTION:
This is a pre-market, monocentre, first-in-human pilot on adult patients with digital nerve defects. Category C clinical trial, medical devices. The study will be performed in Switzerland.

SilkBridge is a biocompatible silk fibroin-based scaffold, which recruits the patients' own cells to remodel or regenerate the nerve, without pre-seeding of the scaffold nor biological/chemical treatments.

SilkBridge will provide surgeons with an implant with unique features, such as easy suturability, full biocompatibility and specific biomimetic properties that enhance cells adhesion and integration of the device with the surrounding tissue.

The study will have a 12 months and 1 week duration per patient, including the follow-up period, and with an expected enrollment period of 15 months.

The study will evaluate 15 adult patients, aged 18-65 years, diagnosed with digital nerve defects (> 5 mm gap) in whom surgical repair may not allow direct suture.

ELIGIBILITY:
Inclusion Criteria:

* male & female patients between 18 and 65 years of age
* a traumatic injury or a post-traumatic neuroma of a digital nerve on the palmar side of the hand, between the metacarpophalangeal joint and the distal interphalangeal joint
* single lesion per finger
* nerve defect of >5mm
* nerve treatment initiated within 24 months after nerve injury
* signed informed consent

Exclusion Criteria:

* disorders known to affect the peripheral nervous system, such as, but not only, diabetes mellitus, chronic heavy alcohol use, or toxic nerve lesions, or any polyneuropathy
* an additional injury that could compromise nerve regeneration
* clinically significant (as defined by the investigator) renal, hepatic, cardiac, endocrine, metabolic, hematologic, autoimmune, or any systemic disease, which may make implementation/interpretation of the protocol or results difficult
* previous conditions of the hand that could affect the healing of the actual nerve injury
* complete amputation injury
* extensive crush injury
* grossly contaminated wound
* receiving immunosuppressive or antineoplastic agents within 30 days prior to the enrolment
* known to be HIV positive
* known pregnant and lactating females
* participated in another clinical investigation using an investigational new drug or device (or in the present study) within 30 days prior to enrolment into this investigation
* uncooperative or unsuitable, e.g. language problems or a suspicion to be unable to attend follow up appointments, for completion of the investigation
* absence of a healthy opposite finger
* suspected allergy to silk
* need of emergency surgery (within 24 hours from injury)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Safety of SilkBridge | 12 months
  Assess type and severity of adverse device effects related to SilkBridge and surgical procedure throughout the follow-up period

SECONDARY OUTCOMES:
Performance - assess at each study visit versus baseline | 12 months
  Sensory recovery after nerve reconstruction by static and moving 2-point discrimination and Semmes-Weinstein monofilament testing Pain evaluation via a visual analog scale (VAS: scale where patient has to specify level of pain by indicating a position along a continuous line between two end-points (0 - 10). 0 indicates no pain while 10 represents the highest level.)
Performance - assess at V5 and at last visit versus opposite control finger | 6 and 12 months
  Sensory recovery by static and moving 2-point discrimination and Semmes-Weinstein monofilament testing
Performance - assess at the last visit | 12 months
  Patient's satisfaction through the Patient Global Impression of Change (PGIC) questionnaire (Patient has to describe the change (if any) in activity limitations, symptoms, emotions and overall quality of life, in relation to its painful condition. 0 value represent no change, 7 a considerable improvement).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Calcagni, MD, Principal Investigator — Klinik für Plastische Chirurgie und Handchirurgie - UniversitätsSpital Zürich
Locations (1):
- Klinik für Plastische Chirurgie und Handchirurgie - UniversitätsSpital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Faroni A, Mobasseri SA, Kingham PJ, Reid AJ. Peripheral nerve regeneration: experimental strategies and future perspectives. Adv Drug Deliv Rev. 2015 Mar;82-83:160-7. doi: 10.1016/j.addr.2014.11.010. Epub 2014 Nov 14. PMID 25446133
- [Background] Konofaos P, Ver Halen JP. Nerve repair by means of tubulization: past, present, future. J Reconstr Microsurg. 2013 Mar;29(3):149-64. doi: 10.1055/s-0032-1333316. Epub 2013 Jan 9. PMID 23303520
- [Background] Wieringa PA, Goncalves de Pinho AR, Micera S, van Wezel RJA, Moroni L. Biomimetic Architectures for Peripheral Nerve Repair: A Review of Biofabrication Strategies. Adv Healthc Mater. 2018 Apr;7(8):e1701164. doi: 10.1002/adhm.201701164. Epub 2018 Jan 19. PMID 29349931
- [Background] Ichihara S, Inada Y, Nakamura T. Artificial nerve tubes and their application for repair of peripheral nerve injury: an update of current concepts. Injury. 2008 Oct;39 Suppl 4:29-39. doi: 10.1016/j.injury.2008.08.029. PMID 18804584
- [Background] Pfister LA, Papaloizos M, Merkle HP, Gander B. Nerve conduits and growth factor delivery in peripheral nerve repair. J Peripher Nerv Syst. 2007 Jun;12(2):65-82. doi: 10.1111/j.1529-8027.2007.00125.x. PMID 17565531
- [Background] Daly W, Yao L, Zeugolis D, Windebank A, Pandit A. A biomaterials approach to peripheral nerve regeneration: bridging the peripheral nerve gap and enhancing functional recovery. J R Soc Interface. 2012 Feb 7;9(67):202-21. doi: 10.1098/rsif.2011.0438. Epub 2011 Nov 16. PMID 22090283
- [Background] Meek MF, Varejao AS, Geuna S. Use of skeletal muscle tissue in peripheral nerve repair: review of the literature. Tissue Eng. 2004 Jul-Aug;10(7-8):1027-36. doi: 10.1089/ten.2004.10.1027. PMID 15363160
- [Background] Vepari C, Kaplan DL. Silk as a Biomaterial. Prog Polym Sci. 2007;32(8-9):991-1007. doi: 10.1016/j.progpolymsci.2007.05.013. PMID 19543442
- [Background] Thurber AE, Omenetto FG, Kaplan DL. In vivo bioresponses to silk proteins. Biomaterials. 2015 Dec;71:145-157. doi: 10.1016/j.biomaterials.2015.08.039. Epub 2015 Aug 20. PMID 26322725
- [Background] De Vita R, Buccheri EM, Pozzi M, Zoccali G. Direct to implant breast reconstruction by using SERI, preliminary report. J Exp Clin Cancer Res. 2014 Nov 25;33(1):78. doi: 10.1186/s13046-014-0078-5. PMID 25422034
- [Background] Lee JH, Lee JS, Kim DK, Park CH, Lee HR. Clinical outcomes of silk patch in acute tympanic membrane perforation. Clin Exp Otorhinolaryngol. 2015 Jun;8(2):117-22. doi: 10.3342/ceo.2015.8.2.117. Epub 2015 May 13. PMID 26045909